CLINICAL TRIAL: NCT02359513
Title: Evaluation of the Efficacy of Serotoninergic Antidepressants in Bulimia Nervosa, According to Brain Serotonin Profile Determined by Positron Emission Tomography With [18F] MPPF - a Multicenter Study
Brief Title: Evaluation of the Efficacy of Serotoninergic Antidepressants in Bulimia Nervosa, According to Brain Serotonin Profile Determined by Positron Emission Tomography With [18F] MPPF.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1408170; 2015-000365-31 (EudraCT Number)
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Bulimia Nervosa
Keywords: bulimia; serotoninergic brain activity; fluoxetine; serotoninergic antidepressant; brain serotonin profile; positon emission tomography
MeSH Terms: conditions — Bulimia Nervosa; Bulimia | interventions — Antidepressive Agents; Fluoxetine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- boulimic (Experimental): Analyse of serotoninergic brain activity (determined by positron emission tomography using [18F]MPPF) from bulimic patients treated with serotoninergic antidepressants during 3 months. The serotoninergic brain activity is measured before adnd after the serotoninergic antidepressant treatment.
  Interventions: Drug: Antidepressants; Drug: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Antidepressants — bulimic patients are treated during 3 months
  Other Names: Fluoxetine
Drug: Positron Emission Tomography (PET) — PET scan using [18F]MPPF is performed before and after (3 months)antidepressant treatment
  Other Names: PET scan

SUMMARY:
Bulimia nervosa (BN) is a serious mental illness characterized by massive food crises followed by anxiety and compensatory behaviours (vomiting more often). Recent data show an increasing prevalence and a serious prognosis, due to excess mortality by suicide but also somatic complications.

Two types of treatments are validated : serotoninergic antidepressants (SSRI) and psychotherapy. Many clinical trials confirm the effectiveness of the SSRI. But many studies also emphasize the important proportion of non-responders to SSRI, few of them analyze the reasons for this non-answer.

To better understand the mode of action of SSRI, we should analyse the serotonergic activity in the central nervous system in bulimia. Recently, specific brain 5HT1A serotonin receptor ligands ([18F] MPPF or [11 C] WAY-100635), were used in positron emission tomography (PET) to characterize the serotonergic abnormalities of bulimic patients. The ligand [18F] MPPF has the feature to be sensitive to the level of endogenous serotonin.

A first pilot study using PET with [18F] MPPF realized between the University Hospital of Saint Etienne and Lyon CERMEP showed a diffuse increase of the binding potential of [18F] MPPF in bulimic patients, suggesting a decrease in serotonin activity.

The brain regions affected were angular gyrus, medial frontal cortex, left insula, cingulate gyrus and orbitofrontal gyrus. These areas are involved in major bulimic symptoms (impulse, taste, instinct, anxiety and satiety). However, we noticed an interindividual heterogeneity of cortical binding of [18F] MPPF.

In front of the heterogeneity in terms of efficacity of SSRI and brain serotoninergic activity, it seems necessary to continues investigations, to determine if there is a link between brain serotonin profile and responding to SSRI in bulimia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Bulimic patients according to DSM-IV TR: minimum 2 bulimic crises (compulsive eating followed by compensatory behavior) / week for 3 weeks
* Patients who signed informed consent to the study
* BMI greater than or equal to 18.5 kg / m²

Exclusion Criteria:

* Against-indication to the SSRI or fluoxetine
* SSRI consumption in the previous three months
* Other addiction (except tobacco, for reasons of feasibility)
* Diagnosis of binge eating disorder or EDNOS (DSM-IV-TR)
* Patients with heart failure
* Against-indication for PET and / or MRI: pacemaker, intracerebral clips, prosthesis made of ferromagnetic material or claustrophobia
* Subjects with suspected pregnancy or in the second half of their menstrual cycle in the absence of oral contraceptives; positive Β-HCG test before the exam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Correlation between [18F]MPPF Binding Potential (BP) and efficacy of antidepressant treatment | 3 months
  Correlation between efficacy of antidepressant treatment quantified by change from the baseline in number of bulimic crises and the change from the baseline in [18F]MPPF BP at 3 months

SECONDARY OUTCOMES:
Correlation between [18F]MPPF Binding Potential (BP) and psychometric scores | 3 months
  Correlation between change from the baseline in [18F]MPPF BP and change from the baseline in psychometric scores at 3 months
Correlation between [18F]MPPF Binding Potential (BP) and initial severity | 3 months
  Correlation between [18F]MPPF Binding Potential (BP) at 3 months and initial (month 0) disease severity quantified by numbers bulimic crises over last 2 weeks before the initial evaluation and psychometric scores at initial evaluation (day 0)
Change from baseline in [18F]MPPF Binding Potential (BP) | 3 months
  Comparison between [18F]MPPF Binding Potential (BP) before antidepressant treatment (day 0) and after antidepressant treatment (month 3)

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan GALUSCA, MD, Principal Investigator — CHU SAINT-ETIENNNE
Locations (4):
- France (4):
  - Groupement Hospitalier Est - HCL, Bron
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No